CLINICAL TRIAL: NCT01940666
Title: Clinical and Biochemical Presentations of Distinctive Types of Biochemical Hyperandrogenism in Premenopausal Taiwanese Women
Brief Title: Presentations of Hyperandrogenic Phenotypes in Taiwanese Women
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ming-I Hsu, Taipei Medical University WanFang Hospital, Taipei Medical University WanFang Hospital
Other Study IDs: WFH-TMU-PCOS-201207025
Record Dates: First submitted 2013-04-05; First posted 2013-09-12 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Hyperandrogenism,; Polycystic Ovary Syndrome,; Metabolic Syndrome,; Insulin Resistance,; Cardiovascular Disease.
Keywords: Hyperandrogenism/; FAI/; Metabolic syndrome/; Adipocytokines/; Insulin resistance.
MeSH Terms: conditions — Hyperandrogenism; Polycystic Ovary Syndrome; Metabolic Syndrome; Insulin Resistance; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Controls: patients who have all androgens (TT, A4, FAI, and DHEA-S) lower than their cut-off values
- Total Testosterone >= 2.39: Patients who have only total testosterone higher than its cut-off value; (TT) >=2.39
- Androstenedione >= 2.99: Patients who have only androstenedione higher than its cut-off value; (A4) >=2.99
- Free Androgen Index >= 6.53: Patients who have only free androgen index higher than its cut-off value; (FAI) >=6.53
- DHEAs >= 181.55: Patients who have only dehyroepiandrosterone sulfate higher than its cut-off value; (DHEA-S)>=181.55

SUMMARY:
STUDY QUESTION: Which of the four abnormally elevated androgen groups (total testosterone [TT], androstenedione [A4], free androgen index [FAI], or dehydroepiandrosterone-sulfate [DHEA-S]) present with an unfavorable metabolic and hormonal profile, appear to be more insulin-resistant and pose additional cardiovascular risk? SUMMARY ANSWER: Subjects with excess free androgen index tend to be obese and face the highest metabolic syndrome risk, adipocytokine alterations, insulin resistance (IR) and cardiovascular risk. The excess TT group presents with a marginal IR risk, while the excess A4 group has the highest antimüllerian hormone (AMH), and may counterbalance obesity; this group and the excess DHEA-S group have a favorable association with IR.

DETAILED DESCRIPTION:
STUDY DESIGN, SIZE, DURATION:A retrospective study in 160 Taiwanese women with HA and 165 women without HA, with medical records reviewed from 2009 up to 2012. The hyperandrogenic women were classified into four groups (TT, A4, FAI, and DHEA-S) according to independent abnormally elevated androgen measures each above its cut-off value, and the groups were compared with each other and with controls.

PARTICIPANTS/MATERIALS, SETTING, METHODS: This study was performed in the Reproductive Endocrinology Clinic at Wan Fang Medical Center in Taipei, Taiwan. Anthropometric, metabolic, endocrine, and IR components as well as lipid accumulation product (LAP) index were compared between the groups. IR was assessed with the following markers: fasting glucose and insulin levels, oral glucose tolerance test, glucose-to-insulin ratio and homeostasis model assessment of IR index (HOMA-IR).

ELIGIBILITY:
Inclusion Criteria:

* Hyperandrogenic women who were classified into four groups:

  * Total testosterone (TT),
  * Androstenedione (A4),
  * Free androgen index (FAI),
  * and Dehydroepiandrosterone sulphate(DHEA-S).
* According to abnormally elevated androgen measures each above its cut-off value, and non hyperandrogenic women (who had all androgens below their cut-off values)

Exclusion Criteria:

* None of the women studied had

  * Hypogonadotropic hypogondism,
  * Hyperprolactinemia,
  * Congenital adrenal hyperplasia,
  * Premature ovarian failure,
  * Androgen-secreting tumors,
  * Cushing's syndrome,
  * or any other endocrine or systemic disease that may affect the reproductive function,
  * or any disorders of the uterus (e.g. Asherman's syndrome and Mullerian genesis) and chromosomal anomalies (e.g. Turner's syndrome).
* In addition, we excluded females who had

  * Experienced menarche less than three years preceding the study start,
  * or who had day 3 FSH > 15 mIU/ml, as well as women with insufficient clinical/biochemical records,
  * and women with ovarian cysts or tumors in an ultrasonographic examination.

Ages: 13 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A retrospective review of the medical records of women who visited the Reproductive Endocrinology Clinic was carried out at the Wan Fang Medical Center at Taipei Medical University from 2009 and up to 2012. A total of 160 Taiwanese women with hyperandrogenism (HA) and 165 women without hyperandrogenism (non-HA) were included in the study.
Sampling Method: Probability Sample
Enrollment: 649 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Clinical and Biochemical Presentations of Distinctive Types of Biochemical Hyperandrogenism in Premenopausal Taiwanese Women | A retrospective study in 160 Taiwanese women with HA and 165 women without HA, with medical records reviewed from January 1, 2009, through July 21, 2012 (up to 3.5 years)
  Androgens (Total Testosterone (TT) (nmol/L), androstenedione (A4)(ng/ml), free androgen index (FAI), and dehydroepiandrosterone sulfate (DHEA-S) (µg/dl ); anthroponmetric components (body mass index (BMI)(Kg/m2) , waist (cm), Waist-to-hip ratio (W/H)); average menstrual interval, antimullerian hormone(AMH)(ng/ml) adiponectin (ng/nl), leptin(ng/ml), adiponectin/leptin (A/L) ratio, and insulin resistance markers( fasting insulin (µIU/ml), glucose-to-insulin ratio (GIR), Homeostasis model assessment insulin resistance (HOMA-IR) Index, Lipid Accumulation Product Index (LAP Index)).

CONTACTS AND LOCATIONS:
Overall Officials: Ming I Hsu, MD, Principal Investigator — WanFang Medical Center at Taipei Medical University
Locations (1):
- WanFang Medical Center at Taipei Medical University, Taipei, Taiwan, Taiwan